CLINICAL TRIAL: NCT06007976
Title: Impact of Variable Treatment Frequencies of Low-Level Laser in Reduce Low-Back Pain
Brief Title: LLLT to Reduce Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Erchonia Corporation (Industry)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-004998
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
Keywords: laser; LLLT; back pain; pain; low back pain
MeSH Terms: conditions — Low Back Pain; Back Pain; Pain

STUDY DESIGN:
Intervention Model Description: All patients will self-select one of four treatment options: 1 week (2 treatment), 2 weeks (4 treatments), 3 weeks (6 treatments) and 4 weeks (8 treatments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- 2 treatment (Experimental): Subjects will receive 2 low-level laser therapy treatments of 20 minutes for low back pain.
  Interventions: Device: Erchonia® Trident
- 4 treatment (Experimental): Subjects will receive 4 low-level laser therapy treatments of 20 minutes over 2 weeks for low back pain.
  Interventions: Device: Erchonia® Trident
- 6 treatment (Experimental): Subjects will receive 6 low-level laser therapy treatments of 20 minutes over 3 weeks for low back pain.
  Interventions: Device: Erchonia® Trident
- 8 treatment (Experimental): Subjects will receive 8 low-level laser therapy treatments of 20 minutes over 4 weeks for low back pain.
  Interventions: Device: Erchonia® Trident

INTERVENTIONS:
Device: Erchonia® Trident — Low-level laser therapy

SUMMARY:
The purpose of this research study is to gather information on the effectiveness of the Trident low-level laser therapy (LLLT) in combination with clinical patient education manuals to reduce lower back pain.

DETAILED DESCRIPTION:
Patients will be administered one of 4 treatment options using the Trident LLLT. The treatment options include 2 treatments, 4 treatments, 6 treatments or 8 treatments. All patients will receive two self-help patient education manuals. Low Back Pain will be compared among all 4 options at the end of week 6.

ELIGIBILITY:
Inclusion Criteria:

* Reporting a primary pain point in lower back.
* Pain intensity reported at baseline must be 4 and above on the Visual Analogue scale (PROMIS Numeric Rating Scale).
* Individual able to participate fully in all aspects of the study and have understood and signed study informed consent.

Exclusion Criteria:

* Have used pain medications or participated in a pain treatment within three days of study enrollment.
* Have an implanted device (including lap band) in the targeted area of Low Level Laser Treatment.
* Have used an investigational drug within 30 days of study enrollment.
* Reports being currently pregnant, lactating, or are of child-bearing potential or are likely to become pregnant during the low level laser treatment phase and are unwilling to use a reliable form of contraception. Acceptable forms of contraception include: Hormonal methods, such as birth control pills, patches, injections, vaginal ring, or implants; Barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm); Intrauterine device (IUD); Total hysterectomy or tubal ligation; Abstinence (no sex).
* Have a history of any major cardiovascular events including heart valve disease, ongoing angina, cardiac arrhythmias, congestive heart failure, acute coronary syndrome, stroke, transient ischemic attack, or peripheral vascular disease.
* Have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, metabolic disease (such as uncontrolled diabetes type 2), active cancer, actively receiving l treatment for cancer or within 1 year of cancer remission.
* Surgical intervention for pain within 1 month prior to enrollment.
* Active infection, wound or other external trauma to the areas to be treated with the laser
* Known photosensitivity disorder.
* Have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Pain Inventory score | Baseline, Week 6
  The PROMIS Numeric Rating Scale v1.0 - Pain Intensity 1a will be used to measure pain intensity on a VAS scale where '0' is no pain and '10' being the worst imaginable pain.
Change in Brief Pain Inventory score | Baseline, Week 24
  The PROMIS Numeric Rating Scale v1.0 - Pain Intensity 1a will be used to measure pain intensity on a VAS scale where '0' is no pain and '10' being the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Mayo Clinic; Ryan T Hurt, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials